CLINICAL TRIAL: NCT01800539
Title: Improving Part C Services and Outcomes for Under-resourced Children With ASD
Brief Title: Improving Services and Outcomes for Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Landa, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00023642
Record Dates: First submitted 2013-02-04; First posted 2013-02-27 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; Early Intervention; Minority
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provider Education Model (PEM) (Experimental): condition wherein providers will receive specially structured training during their typical home visits based by Kennedy Krieger Institute (KKI) staff
  Interventions: Behavioral: Provider Education Model (PEM)
- Treatment-as-Usual (TAU) (No Intervention): condition wherein providers continue with their existing practices

INTERVENTIONS:
Behavioral: Provider Education Model (PEM) — Providers will be trained to use evidence-based practices for early intervention service delivery in the Autism Spectrum Disorder population.
  Arms: Provider Education Model (PEM)

SUMMARY:
Based on the need to characterize and improve early intervention services for minority and under-resourced children with ASD, this study translates a manualized and proven training model to examine its impact on the use of evidence-based practices (EBP) by early intervention providers, and to examine its relationship to child and family outcomes. By highlighting the impact of EBP-focused training on participating providers, children, and families, findings of the proposed study have the potential to effect significant change in the organization and delivery of early intervention services for minority and under-resourced children with ASD.

ELIGIBILITY:
Inclusion Criteria for Providers:

* Providers must be employed by an Infants and Toddlers Program; and
* Serve at least one eligible child with ASD

Inclusion Criteria for Families/Children:

* Children must be between 12 months, 0 days and 35 months, 30 days of age at entry into the study;
* Children must meet criteria on the Autism Diagnostic Observation Schedule (ADOS) for ASD or autism; and
* Caregiver and child must be available for all assessments

Exclusion Criteria for Families/Children:

* Children will be excluded if they are in foster care or wards of the state
* Caregiver must be fluent in speaking and understanding the English language

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Change in Provider Delivery Service Practices | Baseline and 6 months into treatment
  Provider measure

SECONDARY OUTCOMES:
Change in Baseline Mullen Scales of Early Learning | Baseline and 6 months into treatment
  Child measure
Change in Baseline Autism Diagnostic Observation Schedule | Baseline and 6 months into treatment
  Child measure
Change in Caregiver Interaction with Child | Baseline and 6 months into treatment
  Caregiver measure

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States